CLINICAL TRIAL: NCT06422494
Title: The Role of the Adrenergic System in Hypoglycaemia Induced Inflammatory Response in People With Type 1 Diabetes and People Without Type 1 Diabetes-RAID-II
Acronym: RAID-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 115142
Record Dates: First submitted 2024-05-08; First posted 2024-05-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 1; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Inflammation | interventions — Propranolol; Phentolamine

STUDY DESIGN:
Intervention Model Description: Potentially eligible adult ( 16 - 75 years) participants will be recruited through social media, the Radboudumc outpatient clinic and other advertisements. We will recruit a total of 24 individuals, i.e. 12 healthy participants and 12 participants with type 1 diabetes. Participants with type 1 diabetes will be twice ( as there are two investigational days) equipped with a blinded continuous glucose monitoring device (CGM) during the test, which will measure interstitial glucose levels for a total of 10 days.
Who Masked: Participant
Masking Description: Participants will be blinded tot the co-infusion during hypoglycaemia. This will be achieved by similar labelling, with phentolamine having the label infusion A and the propranolol infusion having the label infusion B. When administering saline the 50 milliliter syringes will be filled with saline instead of the solution containing either phentolamine or propranolol. Both saline syringes will still have the labels infusion A and infusion B. The investigators will not be blinded as they will be preparing the adrenergic solutions and the saline solutions. The participants will receive the same amount of millilitres during both infusions, determined by the amount infused during adrenergic blockade. Participants will be block-randomized with blocks of 2 using a randomisation list allocated to receive either the adrenergic blockade or the saline first. The coordinating investigator will have access to this list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants without type 1 diabetes (Active Comparator): The participants without type 1 diabetes
  Interventions: Drug: hyperinsulinaemic hypoglycaemic clamp; Drug: Propranolol Hydrochloride 1 MG/ML; Drug: Phentolamine
- Participants with type 1 diabetes (Active Comparator): Participants with type 1 diabetes
  Interventions: Drug: hyperinsulinaemic hypoglycaemic clamp; Drug: Propranolol Hydrochloride 1 MG/ML; Drug: Phentolamine

INTERVENTIONS:
Drug: hyperinsulinaemic hypoglycaemic clamp — Insulin will be infused at a continuous rate of 60 mU∙m-2 ∙min-1 and glucose 20% will be infused at a variable rate, aiming for stable plasma glucose levels of 5.0 mmol/L. The infusion rate of glucose will be adjusted by plasma glucose levels, measured at 5-minute intervals. After 30 minutes of stable euglycaemia, plasma glucose levels will be allowed to drop gradually to 2.8 mmol/L and will be maintained at this level for 60 minutes. Then, insulin infusion and adrenergic blockade infusions will be stopped. Glucose infusion will be increased and then tapered until stable euglycaemia plasma levels are reached.
Drug: Propranolol Hydrochloride 1 MG/ML — When euglycaemic level of 5.0mmol/L is achieved we will start the adrenergic blockade which will continue throughout euglycaemia and hypoglycaemia. The participants will be administered a bolus of phentolamine of 70µg/kg followed by a dose of 7.0µg/kg/min continuous infusion and a bolus of propranolol of 14µg/kg followed by a dose of 1.4µg/kg/min.
Drug: Phentolamine — When euglycaemic level of 5.0mmol/L is achieved we will start the adrenergic blockade which will continue throughout euglycaemia and hypoglycaemia. The participants will be administered a bolus of phentolamine of 70µg/kg followed by a dose of 7.0µg/kg/min continuous infusion and a bolus of propranolol of 14µg/kg followed by a dose of 1.4µg/kg/min.

SUMMARY:
The goal of this trial is to study the effect that adrenaline has on the immune reaction seen during a low blood sugar. People with type 1 diabetes do not produce their own insulin. The cells in the pancreas that produce insulin are destroyed. People with type 1 diabetes require daily insulin administration. As a consequence of this insulin therapy the blood sugar can dip too low, causing symptoms such as confusion, irritation and tiredness. This is called hypoglycaemia. Hypoglycaemia has been associated with an increased risk for cardiovascular disease such as heart attacks. During hypoglycaemia the immune system is activated. The immune system consists of white blood cells which produce cytokines, these are proteins used to kill pathogens such as bacteria. During hypoglycaemia there are no pathogens but the cytokines are still produced, leading to unwanted damage. A previous study performed by our research group showed that the immune system activation caused by hypoglycaemia is associated with the stress hormone adrenaline. Adrenaline is released by the body in moments of stress such as during running or bungee jumping. Adrenaline is also released by the body during hypoglycaemia to increase the sugar level. Our hypothesis is that adrenaline activates the immune system during hypoglycaemia. Adrenaline acts in the body through two receivers, these are called alpha and beta receptors. These are present on almost all cells in the body especially on the immune cells. With the study we want to study the situation where there is a hypoglycaemia without the adrenaline. We will achieve this by lowering the blood sugar in participants. During the low blood sugar we will administer two drugs, which will attach themselves to the adrenaline receivers, the alpha and beta receptor. With this method we hope to block the adrenaline effects and with that block the immune response caused by adrenaline.

DETAILED DESCRIPTION:
Rationale: Hypoglycaemia has shown to cause a sustained pro-inflammatory response which could promote a pro-atherogenic state and explain the association between hypoglycaemia and cardiovascular events. This pro-inflammatory response has been linked to the adrenaline response to hypoglycaemia. Adrenergic blockade with α and β adrenergic receptor antagonists (ARA) has shown to blunt the leukocyte response after hypoglycaemia induction and adrenaline administration. Whether and to what degree a combined blockade blunts the hypoglycaemia induced pro-inflammatory response is unknown.

Objective: to examine the effect of adrenergic inhibition on the hypoglycaemia induced inflammatory response (e.g. leukocyte phenotype, cytokines, inflammatory proteins) by performing a hyperinsulinaemic hypoglycaemic glucose clamp alongside infusion of α-ARA and β-ARA. Secondary objectives consist of the effect of adrenergic blockade during hypoglycaemia on atherogenic parameters and glucose metrics ( e.g. time in range).

Study design: Intervention study with a cross-over design

Study population: Potentially eligible adult ( 16 - 75 years) participants will be recruited through social media, the Radboudumc outpatient clinic and other advertisements. We will recruit a total of 24 individuals, i.e. 12 healthy participants and 12 participants with type 1 diabetes. Participants with type 1 diabetes will be twice ( as there are two investigational days) equipped with a blinded continuous glucose monitoring device (CGM) during the test, which will measure interstitial glucose levels for a total of 10 days.

Intervention: All participants will undergo a hyperinsulinaemic hypoglycaemic glucose clamp ( nadir 2.8 mmol/L). During the clamp the participants will be randomized to receive an infusion of saline or an infusion of phentolamine and propranolol. This will be done using a cross-over design. The participants will undergo both the saline and adrenergic blockade.

Main study parameters/endpoints: The main study parameter will be the monocyte count after 60 minutes hyperinsulinaemic hypoglycaemic clamp and adrenergic blockade during the clamp.

ELIGIBILITY:
Inclusion Criteria:

* Overall inclusion criteria:

  * Ability to provide written informed consent
  * Body-Mass Index: 18,5-35 kg/m2
  * Age ≥16 years, ≤ 75 years
  * Blood pressure: <140/90 mmHg
  * Non-smoking
  * Electrocardiogram not showing any serious arrythmias (premature ventricular complexes and premature atrial complexes accepted)

Diabetes group specific criteria:

* Insulin treatment according to basal-bolus insulin regimen (injections or insulin pump)
* Duration of diabetes > 1 year
* HbA1c < 100 mmol/mol,

Exclusion Criteria:

* Any event of cardiovascular disease in the past 5 years (e.g. myocardial infarction, stroke, symptomatic peripheral arterial disease)
* Pregnancy or breastfeeding or unwillingness to undertake measures for birth control
* Active epilepsy ( with the need for treatment)
* Allergy for sulphite
* Active asthma with use of β2-bronchodilators or obstructive lung disease
* Current treatment with Alpha- or beta-blockers (e.g. doxazosin, propranolol)
* History of clinical significant Arrhythmias
* Use of immune-modifying drugs or antibiotics
* Use of antidepressants ( Including monoamine oxidase inhibitors, tricyclic antidepressants and serotonin-reuptake inhibitors)
* Use of antipsychotics
* Use of statins with the inability to stop statins >2 weeks before the investigational day.
* Proliferative retinopathy
* Nephropathy with an estimated glomerular filtration rate (by Chronic Kidney Disease Epidemiology Collaboration equation, CKD-EPI) ˂60ml/min/1.73m2

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — We aim to match our participants with each other to have comparable groups. So we aim to have the same amount of males and females.
Enrollment: 24 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Monocyte count after 60 minutes of hypoglycaemia and adrenergic blockade | After 60 minutes of hypoglycaemia and adrenergic blockade
  The number of monocytes following 60 minutes hypoglycaemia and adrenergic blockade compared to baseline. Adrenergic blockade using Phentolamine and Propranolol intravenously. Expressed in 10^3/µl measured using a sysmex machine.

SECONDARY OUTCOMES:
Leukocyte count at the time points | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia, +1 day, +3 days and 1 week after of hypoglycaemia
  Leukocyte count at the time points 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia, +1 day, +3 days and 1 week after of hypoglycaemia (e.g. Monocytes, granulocytes, lymphocytes).
Ex vivo production of pro- and anti-inflammatory cytokines and chemokines | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia, +1 day, +3 days and 1 week after of hypoglycaemia
  Ex vivo production of pro- and anti-inflammatory cytokines and chemokines after ex vivo stimulation of isolated leukocytes, including Tumor necrosis factor-α, Interleukin-6, Interleukin-10 and Interleukin-1β, 1β
92 circulating inflammatory proteins | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  92 circulating inflammatory proteins using Olink Proteomics inflammation panel
Inflammatory plasma protein ( e.g. high-sensitive crp) | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Inflammatory plasma protein using ELISA,(e.g high sensitive-crp)
Atherogenic parameters | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Atherogenic parameters using ELISA including but not limited to, vascular endothelial cell adhesion molecule-1, vascular endothelial cell adhesion molecule-1, E-Selectin, P-selectin, Plasminogen activator inhibitor-1, Plasma Endothelin
Plasma levels of hormones | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Plasma levels of hormones ( Cortisol, insulin, glucagon, growth-hormone, adrenaline, noradrenaline)
Amount of hypoglycaemic events measured by the blinded continuous glucose monitor | During the full study, 3 days before and 7 days after each investigational day
  Amount of events
Variability measured by the blinded continuous glucose monitor | During the full study, 3 days before and 7 days after each investigational day
  Variability of glucose expressed as a standard deviation of the mean glucose
Average glucose measured by the blinded continuous glucose monitor | During the full study, 3 days before and 7 days after each investigational day
  Average glucose during the 10 days of measuring expressed as mmol/L
Time in range measured by the blinded continuous glucose monitor | During the full study, 3 days before and 7 days after each investigational day
  Amount of time that glucose is between 3.8 and 10 mmol/L expressed as a percentage
Amount of plasma glycerol | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Amount of plasma glycerol during and after hypoglycaemia
Amount of Non-esterified fatty acids | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Amount of Non-esterified fatty acids (NEFAs) during and after hypoglycaemia
Untargeted metabolomics profiling | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Measuring a panel of amino acids
Gene expression changes in leukocytes | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Gene expression changes in leukocytes (e.g. using RNA sequencing, quantitative PCR)
Epigenetic changes in leukocytes | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Epigenetic changes in leukocytes (e.g. using Assay for Transposase- Accessible Chromatin using sequencing (ATACseq), DNA methylation analysis)
Functional changes in monocytes | 0, 30 minutes after euglycaemia, 60 minutes during hypoglycaemia
  Functional changes in monocytes (e.g. using adhesion assays, differentiation experiments)
Adrenergic symptoms assessed using the validated Edinburgh Hypoglycaemia Score | 0, 30 minutes after euglycaemia, 30 minutes and 60 minutes during hypoglycaemia
Hypoglycaemia awareness using the modified Clarke score | At screening

OTHER OUTCOMES:
HbA1c expressed in mmol/L | At screening
Serum creatinine for kidney function expressed in umol/L | Once at the screening at least 1 week before the hypoglycaemia
Vitals ( blood pressure and heart rate) | At both investigational days, every 15 minutes during each investigational day for a total of 8 hours.
  Measured by automatic sphygmomanometer
Body mass index | Once at the screening at least 1 week before the hypoglycaemia
  Using length and weight expressed in kg/m^2
Age | Once at the screening at least 1 week before the hypoglycaemia
Sex | Once at the screening at least 1 week before the hypoglycaemia
  Male or female
Duration of diabetes ( years) | Once at the screening at least 1 week before the hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Cees Tack, MD, PhD, Principal Investigator — Radboud University Medical Center (Radboudumc)
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will share the study protocol using a data repository accessible through the research team on demand. Starting around 6 months after publication.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: The coordinating researcher will review access requests. Seeing as the data are all anonymized access will be granted for additional research in the field of inflammation or diabetes.